CLINICAL TRIAL: NCT00125749
Title: Vaccination of Patients With Stage IV Melanoma With Dendritic Cells Generated Ex Vivo From Monocytes and Loaded With Heat Treated Killed Allogeneic Melanoma Cells
Brief Title: Vaccination of Patients With Stage IV Melanoma With Dendritic Cells
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Collaborators: Mary Crowley Medical Research Center (Other); ODC Therapy (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 005-065-02
Record Dates: First submitted 2005-08-01; First posted 2005-08-02 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2017-06

CONDITIONS: Melanoma; Neoplasm Metastasis
Keywords: Dendritic; Vaccine; Melanoma; Stage IV metastatic melanoma
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Dendritic cell vaccination — Autologous Dendritic Cells Derived from PBMC, Cultured with Cytokines, Pulsed Ex Vivo with Irradiated Allogeneic (Colo 829) Melanoma Cells

SUMMARY:
The purpose of this study is to test a novel dendritic cell (DC) vaccine in patients with Stage IV melanoma.

DETAILED DESCRIPTION:
A novel dendritic cell vaccine has been developed at the Baylor Institute for Immunology Research (BIIR). Pre-clinical studies have found that this dendritic cell vaccine is more efficient in inducing a tumor specific immunity than other dendritic cell vaccines. Further studies in the BIIR have been done with dendritic cells that were loaded with killed melanoma cells from a melanoma cell line treated with heat before loading. Both studies have shown that DCs manufactured in this novel way were more efficient in priming the melanoma specific CD8+ cells. Thus, the strategy for this clinical trial will be to test recent laboratory findings in the clinical setting. An additional objective of the study will be to determine the effectiveness of a frozen vaccine product which differs from previous vaccines that were manufactured "fresh".

This clinical trial will evaluate the novel dendritic cell vaccine in patients with Stage IV melanoma. The trial will accrue a total of 30 subjects. The primary goal of this trial will be to test the safety/tolerability/feasibility of the vaccine preparation and the rate of objective clinical response. A 15% objective response rate will be accepted in patients who have failed previous therapy with IL-2 and/or dacarbazine (DTIC) and/or temozolomide which are standard treatments for patients with malignant melanoma.

Each subject will be given 7 initial injections in a fixed dose amount. The first 4 doses will be given at 2-week intervals (Weeks 0, 2, 4 and 6); the last 3 doses will be given at 4-week intervals (Weeks 10, 14, and 18). Those patients who exhibit stable disease, partial response or complete response after 7 injections will be given 4 more vaccinations. Each of these additional 4 vaccinations will be given 3 months apart (Weeks 36, 48, 72 and 96). Scans and re-staging tests will be performed at scheduled intervals throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Stage M1a, M1b, M1c biopsy proven metastatic melanoma
* Failure of at least one prior chemotherapy regimen of DTIC and/or temozolomide with/without interleukin-2 (IL-2).
* Karnofsky performance status greater than/equal to 80%.
* Measurable metastatic lesions by physical exam or scans.
* Acceptable CBC and blood chemistry results
* Adequate renal function.
* Written informed consent.

Exclusion Criteria:

* Patients who have received more than 8 cycles of chemotherapy for metastatic melanoma.
* Patients who have received chemotherapy less than 4 weeks before beginning the trial.
* Patients who have received interferon (IFN) alpha-2b or granulocyte-monocyte colony-stimulating factor (GM-CSF) less than 4 weeks before beginning the trial.
* Patients who have received high-dose IL-2 less than 4 weeks before beginning the trial.
* Patients with a history of central nervous system (CNS) metastatic melanoma.
* More than 5 hepatic lesions or any hepatic lesion larger than 5 cm.
* Baseline serum LDH greater than 4 times the upper limit of normal.
* Patients who are HIV positive.
* Patients who are pregnant.
* Patients who have received corticosteroids or other agents less than 4 weeks before beginning the trial.
* Patients with asthma, angina pectoris or congestive heart failure.
* Patients with autoimmune diseases such as lupus erythematosus, rheumatoid arthritis or thyroiditis.
* Patients with active infections including viral hepatitis.
* Patients with a history of any other neoplastic disease less than 5 years ago (carcinomas in situ of the cervix and basal/squamous cell carcinomas of the skin, however, can be admitted to the study).

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-07; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of the novel DC vaccination product in human subjects | 3 years
Feasibility of a novel approach to DC manufacture | 3 years
Objective clinical responses | 3 years

SECONDARY OUTCOMES:
Immunogenicity of frozen DC vaccinations | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Anna Karolina Palucka, MD, PhD, Study Director — Baylor Institute for Immunology Research: Baylor University Medical Center
Locations (1):
- Mary Crowley Medical Research Center: Baylor University Medical Center, Dallas, Texas, United States

REFERENCES:
- See also: Click here for more information about this study. — http://www.baylorhealth.com/AdvancingMedicine/GetInvolved/Pages/ResearchStudies.aspx